CLINICAL TRIAL: NCT01510548
Title: Adalimumab (Anti TNF Alfa) in the Management of Acute Lumbar Disc Prolapses - a One Year, Randomized, Placebo Controlled, Double Blind, Single Center Trial
Brief Title: ADALISKIAS: Adalimumab for Acute Disc Prolapse
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, olavi airaksinen, MD, PhD Ass Proff, Head of the Department of Rehabilitation, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM53
Record Dates: First submitted 2012-01-02; First posted 2012-01-16 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Disc Prolapse; Pain
Keywords: Disc prolapse; Pain; Disability
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain | interventions — Biological Products; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adalimumab 20 mg per week (Active Comparator): Patient will get at double blind situation adalimumab 20 mg every week (six injections) injections
  Interventions: Biological: Adalimumab injections for acute disc prolapse patients
- Adalimumab 40 mg per week (Active Comparator): Patient will get at double blind situation adalimumab 40 mg per week injections
  Interventions: Biological: Adalimumab injections for acute disc prolapse patients
- placebo arm (Placebo Comparator): Patient will get at double blind situation placebo (= NaCl liquid solution, absolutely same color as the active drug) injections one per week during six weeks - same as the adalimumab arms
  Interventions: Biological: Adalimumab injections for acute disc prolapse patients

INTERVENTIONS:
Biological: Adalimumab injections for acute disc prolapse patients — see the study protocol. Three arms, which two of them included active medication and one will be placebo( NaCl solution) in controlled double blind setting.
  Other Names: Biologic Drugs for ischias; Humira for ischias

SUMMARY:
Aims:

To study the efficacy and safety of adalimumab versus placebo in the treatment of acute disc prolapse will be will be compared up to 12 months after the start of study drug treatment.

Study type:

A one year,randomized, placebo controlled double blind single center trial.

Patients and study drug treatment:

The study population consist of 99 patients with sciatica caused by herniated disc prolapse.

The study has 3 arms: 33 patients randomized to adalimumab 40mg every week, 33 patients randomized to adalimumab 40mg every other week, and 33 patients randomized to placebo. Study drug treatment period will be six weeks.

Methods:

Clinical evaluation, global assessments and Oswestry Disability Score and visual analog scale (VAS) will be used as the evaluation of clinical results with the disc prolapse patients confirmed by Magnetic Resonance Imaging. Health related quality of life will be assessed by 15-D questionnaire. Safety will be evaluated by medical examinations, adverse events (AE) collection and laboratory measurements throughout the study period.

DETAILED DESCRIPTION:
Aims of this study:

TNF alpha is believed to have a major role in the pathogenesis of sciatica. The efficacy and safety of adalimumab versus placebo in the treatment of acute disc prolapse will be will be compared up to 12 months after the start of study drug treatment. Primary objective of the study is to evaluate the clinical functionality of the patients with Oswestry Disability Score and VAS (leg and back pain) at the end of study drug treatment at week 6. Secondary objectives are to compare the need of operative treatment, sick leave days, pain killer consumption and quality of life between the two study groups up to 12 months after the start of study drug treatment.

Patients and study drug treatment:

The study population consist of 99 patients with sciatica caused by herniated disc prolapse. The patients will be randomized to 3 arms: 33 patients to adalimumab 40mg every week, 33 patients to adalimumab 40mg every other week, and 33 patients to placebo. Study drug treatment period will be six weeks.

The study population will be collected from the patient population with severe sciatica symptoms sent to Spine Unit of Department of Physical and Rehabilitation Medicine in Kuopio University Hospital. The patient information will be given orally by investigators at the first visit and also patient information letter will be given. The informed consent will be signed by the patient and the investigator before any study related procedures. Patient will receive a copy of the written information and signed informed consent form. The patient has the right to discontinue his participation at any time without giving any reason.

The randomisation will be made in groups taken in count the level of disc prolapse and and sex. In emergency cases the randomisation will be opened with the decision of investigator. Each patient require 8 site visits. At the baseline visit (visit 0) the patient history and exclusion and inclusion criteria will be checked and MRI will be done. At visit 1 Visual Analogue Scale, Oswestry disability index and Quality of Life Questionnaire (15-D) and clinical examination of patients will be carried out. In case the MRI is already available at baseline visit, the visit can be combined with visit 1. At the follow up visits (1 week, 2 weeks, 4 weeks, 3 months, 6 months and 12 months after the first injection) Visual Analogue Scale, Oswestry disability index and Quality of Life Questionnaire (15-D), Patients and Physicians Global Assessments and clinical examination of patients will be carried out and the Adverse Events are recorded. If the the study medication do not help the sciatica symptoms enough, disc surgery will be evaluated with decision of investigator and neurosurgeon or orthopaedic surgeon at visit of 6 weeks. With very severe symptoms and signs, major neurological signs or intolerable pain the surgery will be evaluated in any phase of study (see rescue medication).

The patient data will be collected to CRF and source data to patient records, where also sick leave days and the use of pain medication will be collected during each site visit. Patient medication and history will be collected at visit 1. The Adverse Events will be evaluated at each visit and recorded to patient records and CRF.

This study is investigator based study and will be carried out on spine center at the Department of Physical and Rehabilitation Medicine in Kuopio University Hospital. The laboratory and imaging studies will be carried out in the Departments of Clinical Chemistry and Radiology. If the surgery is needed the Department of Neurosurgery and Orthopedics will be asked to work. The Abbott Laboratories Ltd will provide the study medication. Adalimumab is registered in Finland for Rheumatoid Arthritis. The study medication will be given at the site visit by investigator. Injections for week 3 and 5 will be administered by the study subject at home.

Efficacy Assessments:

To confirm the clinical diagnosis of sciatica Magnetic Resonance Imaging using Siemens Avant 1.5 T clinical scanner (Siemens, Erlangen, Germany) will be used. Neural compromise will be assessed according to the system of Pfirrmann et al. from grade 0 (no compromise, normal) to Grade 1 (contact), Grade 2 (deviation) and Grade 3 (compression).

Subjective disability will be measured by the Oswestry Disability Index (0-100%), where 0% represents no disability and 100 % extreme difficult disability.

Pain experience will be measured with self-administered visual analogue scale VAS (range 0-100 mm). It has proved to be a valid index of experimental, clinical and chronic pain.

Patients and physicians Global Assessment will be used as the clinical evaluation of treatment.

Quality of life will be assessed by Finnish 15-D questionnaire

Safety Assessments:

At screening the patients must be evaluated for active and latent TB infections by using PPD and chest x-ray (if not available from previous 3 months prior to screening) and a detailed review of the subjects medical history. Also at screening T SPOT-TB test will be taken.

All patients who receive study drug will be included to the safety analysis. Safety follow-up will continue until 70 days after the last study drug injection. Safety will be assessed by AE collection, physical examination, vital signs and laboratory parameters throughout the study period. Safety laboratory parameters (full blood count, ALT, AST, CRP, ESR) will be evaluated at baseline and at the end of study drug treatment on week 6. Adverse Events will be reported to the local Ethics Committee and National Agency of Medicine according to the regulation 2/2004 Clinical Medicinal Trials on Humans.

Statistical review:

Sample size:

The planned sample size of 33 in each arm is projected to provide 80% power to detect a mean difference of 25 in leg pain VAS at 6 weeks at a two-sided alpha level of 0.0125, assuming that the standard deviation is 20. For Oswestry Disability Index (ODI) 33 patients in each arm, would provide 80% power to detect a mean difference of 16 in ODI score at a two-sided alpha level of 0.0125, assuming a standard deviation of 13. Alpha-level of 0.0125 was selected to correct the multiple testing caused by two primary end-point variables and two comparisons for each variable, placebo versus the two different doses of active treatment. The sample size calculation is based on normality assumption; however the final analysis will be performed using non-parametric method. However the use of baseline value as covariate in the analysis should compensate the lost power due to the use of distribution free-method.

Statistical analysis of the primary end-points:

The aim of the study is to demonstrate the efficacy of adalimumab versus placebo by means of Oswestry Disability Index and Leg Pain VAS at week 6. To maintain the overall 5% significance level of the primary end-points, Bonferroni adjustment will be applied, i.e. in the four significance tests applied to the primary hypothesis; p-value should be below 0.0125 to be considered as statistically significant.

As a primary analysis method, non-parametric analysis of covariance with baseline value as a covariate will be applied to ODI and Leg Pain VAS at week 6 separately for adalimumab 40 mg every week versus placebo and adalimumab 40 mg every other week versus placebo. Intent-to-treat population will be used in the primary analysis.

All patient data will be evaluated by intent-to-treat principle.

For the secondary end-points Bonferroni adjustment will be applied on end-point level.

Rescue medication:

Rescue medication will be arranged in case of lack of efficacy at the discretion of the investigator. If cauda equine symptoms or signs of large neurological defects will occur surgery will be performed. Also if the medication is considered a failure by the investigator's clinical judgment the patients will have the opportunity to be evaluated for disc surgery.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over 18 years of age
* Able and willing to give written informed consent
* Acute or subacute (no more than 2 months) clinical sciatica symptoms caused by herniated disc prolapse confirmed by Magnetic Resonance Imaging (MRI).
* Oswestry Disability Score at least 16% at entry.
* VAS (leg and back pain) at least 40 mm at entry.
* Able and willing to self-administer s.c. injections or have available a suitable person to administer s.c. injections.
* A negative pregnancy test (serum HCG) for women of childbearing potential prior to start of study treatment.

Exclusion criteria:

* Prior treatment with any investigational agent within 30 days, or five half lives of the product whichever is longer.
* Prior treatment with infliximab or etanercept.
* History of chronic back pain.
* Previously operated disc prolapse or other spinal column operation
* Uncontrolled diabetes, unstable ischemic heart disease, congestive heart failure (NYHA III-IV), recent stroke (within three months), chronic leg ulcer and any other condition (e.g. indwelling urinary catheter) which, in the opinion of the investigator, would put the subject at risk by participation in the protocol.
* History of cancer or malignant lymphoproliferative disease other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.
* Positive serology for hepatitis B or C indicating active infection.
* History of positive HIV status.
* Persistent or recurrent infections or severe infections requiring hospitalization or treatment with i.v. antibiotics within 30 days, or oral antibiotics within 14 days prior to enrollment.
* Previous diagnosis or signs highly indicative of central nervous system demyelinating diseases (e.g. optic neuritis, ataxia, apraxia).
* History of active tuberculosis, histoplasmosis or listeriosis.
* Female subjects who are pregnant or breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-03; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Pain | one year
  As primary endpoint the functionality of the patients measured by Oswestry Disability Score and VAS (leg and back pain) will be evaluated and the proportion of patients in each group for the need of surgery at week 6 at the end of the study drug injections.

SECONDARY OUTCOMES:
need for operative treatment and functional status = proportion of patients operated after one year | one year
  As secondary endpoints functionality of the patient, need of operative treatment, sick leave days and pain killer consumption will be evaluated at week 1, 2, 4 and 6, 3 months, 6 months and 12 months 1 year after the start of study treatment.
safety in general | During one year follow up.
  All patients who receive study medication will be included to the safety analysis.
  Blood tests before and after administration will be analysed. Vital signs and clinical examination will be recorded on each visits All adverse and serious adverse events will be evaluated in connection to study medication during the follow-up time.

CONTACTS AND LOCATIONS:
Overall Officials: Olavi Airaksinen, MD, Principal Investigator — MD, Head of Department of PRM
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

REFERENCES:
- [Background] Cooper RG, Freemont AJ. TNF-alpha blockade for herniated intervertebral disc-induced sciatica: a way forward at last? Rheumatology (Oxford). 2004 Feb;43(2):119-21. doi: 10.1093/rheumatology/keh013. Epub 2003 Sep 16. No abstract available. PMID 13130150
- [Background] Cuellar MJ, Montesano XP, Carstens E. Role of TNF-alpha in sensitization of nociceptive dorsal horn neurons induced by application of nucleus pulposus to L5 dorsal root ganglion in rats. Pain. 2004 Aug;110(3):578-587. doi: 10.1016/j.pain.2004.03.029. PMID 15288398
- [Background] Genevay S, Stingelin S, Gabay C. Efficacy of etanercept in the treatment of acute, severe sciatica: a pilot study. Ann Rheum Dis. 2004 Sep;63(9):1120-3. doi: 10.1136/ard.2003.016451. Epub 2004 Apr 28. PMID 15115710